CLINICAL TRIAL: NCT01198067
Title: Phase I Study of Pomalidomide in Relapsed or Refractory Waldenstrom Macroglobulinemia
Brief Title: Pomalidomide in Treating Patients With Relapsed or Refractory Waldenstrom Macroglobulinemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: <75% participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0972; NCI-2012-01882 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2010-02076; 2009-0972 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Waldenstrom Macroglobulinemia; Refractory Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pomalidomide) (Experimental): Patients receive pomalidomide PO on days 1-28 or 1-21. Courses repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase I trial studies the side effects and best dose of pomalidomide in treating patients with Waldenstrom macroglobulinemia that has returned after a period of improvement (relapsed) or does not respond to treatment (refractory). Pomalidomide may stimulate the immune system in different ways and stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of pomalidomide in patients with relapsed or refractory Waldenstrom macroglobulinemia.

SECONDARY OBJECTIVES:

I. To evaluate the safety and toxicity profile of pomalidomide in patients with relapsed or refractory Waldenstrom macroglobulinemia.

II. To evaluate the efficacy of pomalidomide in patients with relapsed or refractory Waldenstrom macroglobulinemia.

OUTLINE: This is a dose-escalation study.

Patients receive pomalidomide orally (PO) on days 1-28 or 1-21. Courses repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Waldenstrom's macroglobulinemia that has relapsed and/or is refractory to at least one prior line of therapy
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at study entry
* Serum creatinine =< 2.0 mg/dL
* Creatinine clearance >= 45 ml/min
* Total bilirubin =< 3 x upper limit of normal (ULN) or direct bilirubin =< 2 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x ULN
* Platelet count >= 20 K/microL
* Absolute neutrophil count >= 500 K/microL
* Disease free of prior malignancies for >= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 to 14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to practice complete abstinence or agree use a latex condom during sexual contact with a FCBP while participating in the study, during dose interruptions and for at least 90 days following study drug discontinuation, even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Able to take aspirin (325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use therapeutic dose warfarin or low molecular weight heparin)
* All study participants must be registered into the mandatory POMALYST REMS program, and be willing and able to comply with the requirements of the POMALYST REMS program

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females; (lactating females must agree not to breast feed while taking pomalidomide or for 28 days after stopping pomalidomide)
* Any medical or psychiatric condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study, or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy within 28 days of the first dose of study drug
* Known hypersensitivity to thalidomide or lenalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of pomalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known positive for human immunodeficiency virus (HIV) or acute hepatitis A or acute or chronic active hepatitis B or C
* Grade > 2 peripheral neuropathy
* Neutrophil count < 1000 K/microL and/or
* Platelet count < 100 K/microL unless infiltration by Waldenström's macroglobulinemia equals or exceed 60% of bone marrow cellularity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-10-06 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheeba K Thomas, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient Eligibility:Waldenstrom relapsed,>/18 - years old,ECOG <~2,Labs NCS,no prior cancers,females not preganant,~1> line(s) prior therapy, no therapy in 4 weeks. Excluded:pregnant, breast-feeding, serious diagnosis,chemotherapy reaction,prior pomalidomide,HIV/ Hepatitis A-C +,concurrent chemotherapy,grade~>2 neuropathy,andANC count <~1000K/ul.
Pre-assignment Details: Six patients were screen failures; did not meet inclusion criteria. Original study design included Arms with assignment to increasing dose escalation including 3 and 4mg Pomolidomide Arms/Cohorts; however, safety concerns early on regarding Dose Limiting Toxicities for 2mg Cohort compelled omitting the 3 and 4mg Arms/Cohorts.
Groups:
- Cohort 2: 2mg Pomolidomide per day per Cycle (Cycle = 28 days)
- Cohort 3: 1mg Pomolidomide per day per Cycle (Cycle = 28 days)
Period: Overall Study
Arm/Group | Cohort 2 | Cohort 3
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10) | 66 (11) | 66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing MTD
Description: Maximum Tolerated Dose
Time Frame: Participants Experiencing Study Medication Maximum Tolerated Dose through Study Completion (Avg. 1 Year)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 6
Participants | 1 | 5

2. Secondary Outcome: Cycles Completed
Description: Length of Treatment
Time Frame: Study Completion (Avg. 1 Year)
Measure: Median (Full Range); unit: Number of Cycles
Arm/Group | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 6
Number of Cycles | 2 [1 to 2] | 7 [4 to 12]

3. Secondary Outcome: Changes in Waldestrom Biomarkers
Description: Average Paraprotein1 gm/dL Change Cycle 1 thru Study
Time Frame: Through Study Completion (Avg. 1 Year)
Measure: Mean (Standard Deviation); unit: Paraprotein #1 gm/dL
Arm/Group | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 6
Paraprotein #1 gm/dL | 0.3 (.1) | 1.4 (.7)

4. Secondary Outcome: Changes in Waldestrom Biomarkers
Description: Average Reduction in IgM Protein mg/dL from Cycle 1 thru Study
Time Frame: Through Study Completion (Avg. 1 Year)
Measure: Mean (Standard Deviation); unit: IgM Protein mg/dL
Arm/Group | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 6
IgM Protein mg/dL | 493 (955) | 1252 (2011)

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected through Study Completion (Avg. 1 Year)
Description: Toxicity graded using NCI Common Terminology Criteria for Adverse Events, v3.0 Nonheme Pomalidomide dose limiting toxicity gr 3 ~>except gr3> fatigue, nausea/vomiting, or nonheme abnormal labs resolving to gr1 / baseline 14 days 1st dose. Hematologic toxicity defined as gr4 neutropenia lasting > 14 days, febrile neutropenia, thrombocytopenia (plt #< 25k) > 14 days. All AEs recorded from study entry/first dose-30 days after last dose and/or AE resolution:1/1/2011 to 6/7/2022.
Arm/Group | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2 (N=3) | Cohort 3 (N=6)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Infection (Knee) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Caudia Equina Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2 (N=3) | Cohort 3 (N=6)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Allergy/Immunology (Other) - Allergic Sinusitis (General disorders) | 1 (1) | 1 (1)
Allergy/Immunology (Other) - Lidocaine (General disorders) | 0 (0) | 1 (1)
Allergy/Immunology (Other) - Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anxiety (Nervous system disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bruising (Vascular disorders) | 0 (0) | 1 (1)
Bruising - Injury / Laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Conjunctival disorder (General disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constitutional Symptoms (Other) - Pelvic Cystic Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 1 (4) | 0 (0)
Depression (Nervous system disorders) | 0 (0) | 1 (1)
Dermatology/Skin (Other) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatology/Skin (Other) - Injury / Laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (10)
Dermatology/Skin (Other) - non-malignant growths (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatology/Skin (Other) - Rash NOS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology/Skin (Other) - Rash: Erithematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatology/Skin (Other) - SCC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatology/Skin (Other)- non-malignant skin cancer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 4 (5)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Dry eye syndrome (General disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Edema limbs (Musculoskeletal and connective tissue disorders) | 2 (7) | 4 (5)
Eye pain (General disorders) | 0 (0) | 1 (2)
Eyelid function disorder - Eyelid edema (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (8) | 6 (14)
Fever (General disorders) | 1 (1) | 1 (5)
Gastrointestinal (Other) - Colorectal polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal (Other) - GERD (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival infection (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2)
Hemoglobin decreased (Investigations) | 0 (0) | 5 (8)
Hypertension (General disorders) | 0 (0) | 2 (2)
Infection - COVID + (Infections and infestations) | 0 (0) | 1 (1)
Infection - Human Rhinovirus (Infections and infestations) | 0 (0) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint infection (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Laryngeal inflamation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphatics (Other) - Left axillary nodule (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Metabolic/Laboratory (Other) - Anemia (Investigations) | 1 (1) | 0 (0)
Metabolic/Laboratory (Other) - Hypercapnia (Investigations) | 3 (3) | 1 (2)
Metabolic/Laboratory (Other) - Hyperglycemia (Investigations) | 0 (0) | 1 (1)
Metabolic/Laboratory (Other) - Hypomagnesemia (Investigations) | 0 (0) | 1 (1)
Metabolic/Laboratory (Other) - Hypophosphatemia (Investigations) | 0 (0) | 1 (1)
Metabolic/Laboratory (Other) - Lymphocyte Abs increased (Investigations) | 0 (0) | 1 (1)
Metabolic/Laboratory (Other) - Vitamin D defficiency (Investigations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1)
Musculoskeletal (Other) - Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal (Other) - Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal (Other) - muscle aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal (Other) - Pulled muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3)
Nail infection (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (5)
Neurology (Other) - Drowsiness (Nervous system disorders) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (2) | 2 (6)
Night Sweats (General disorders) | 0 (0) | 1 (1)
Ocular/Visual (Other) - Blurred Vision (General disorders) | 0 (0) | 1 (1)
Ocular/Visual (Other) - Dysfunctional Tear Syndrome (General disorders) | 0 (0) | 1 (1)
Ocular/Visual (Other) - Edema Lids (General disorders) | 0 (0) | 1 (1)
Ocular/Visual (Other) - Increased Eye Pressure (General disorders) | 0 (0) | 1 (1)
Ocular/Visual (Other) - Irritated Eyes (General disorders) | 0 (0) | 1 (1)
Ocular/Visual (Other) - Ocular Conjunctive Hemmorhage (General disorders) | 1 (1) | 1 (1)
Ocular/Visual (Other) - Watery eyes (General disorders) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Otitis media (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain (Other) (General disorders) | 0 (0) | 1 (1)
Pain (Other) - L Thigh (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (General disorders) | 0 (0) | 5 (9)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pulmonary (Other) - Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (5) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rhinitis infective (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Serum magnesium decreased (Investigations) | 0 (0) | 1 (2)
Serum phosphate decreased (Investigations) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Injury / Laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating (General disorders) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Specify, Other) - SCC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vascular (Other) (Vascular disorders) | 0 (0) | 0 (0)
Vision blurred (General disorders) | 1 (1) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (4)
Watering eyes (General disorders) | 0 (0) | 2 (2)
Wound infection - Injury / Laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wound infection - Injury / Laceration / Infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-02-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT01198067/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT01198067/ICF_001.pdf